CLINICAL TRIAL: NCT03909269
Title: Markers for Glycaemic Control and Continuous Glucose Monitoring in Persons With Type 2 Diabetes on Chronic Haemodialysis
Brief Title: Glycaemic Markers in Persons With Type 2 Diabetes on Haemodialysis
Acronym: GLYCOHEMO
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, DMSc, Head of Nephrology, Rigshospitalet, Denmark
Other Study IDs: GLYCOHEMO
Record Dates: First submitted 2019-03-29; First posted 2019-04-09 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Nephropathy Type 2; Type2 Diabetes
Keywords: HbA1c; Glycated albumin; Fructosamine; Continuous glucose monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for both immediately analyses (basic lab data) and later analyses (glycated albumin, fructosamine, HbA1c for immunoassay) and stored for 10 years whereafter they will be destroyed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Haemodialysis and type 2 diabetes: On chronic haemodialysis and type 2 diabetes
  Interventions: Device: Continuous glucose monitoring; Diagnostic Test: Glycaemic markers; Radiation: Erythrocyte life span; Device: Carbon monoxide (CO)-rebreathing method
- Control group: Type 2 diabetes and with eGFR above 60ml/min
  Interventions: Device: Continuous glucose monitoring; Diagnostic Test: Glycaemic markers; Radiation: Erythrocyte life span

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring five times over 17 weeks
Diagnostic Test: Glycaemic markers — Measurement of HbA1c by immunoassay (Roche) and chromatography (TOSOH), including glycated albumin and fructosamine.
Radiation: Erythrocyte life span — Erythrocyte life span measured by Crom-51 labelling over 4 weeks
Device: Carbon monoxide (CO)-rebreathing method — Measurement of total blood volume, plasma volume and erythrocyte volume
  Groups: Haemodialysis and type 2 diabetes

SUMMARY:
To investigate the correlation between the mean glucose concentration measured by continuous glucose monitoring (CGM) and the estimated mean blood glucose from glycated haemoglobin A1c (HbA1c) in persons with type 2 diabetes and on chronic haemodialysis. Furthermore, the aim is to compare CGM and HbA1c with glycated albumin and fructosamine.

DETAILED DESCRIPTION:
Background:

In persons with diabetes, glycated haemoglobin A1c (HbA1c) is used as a retrospective measurement of the patient's estimated mean blood glucose over the past 3 months. HbA1c forms in a non-enzymatic pathway when haemoglobin is exposed to blood glucose. The normal range of HbA1c and the correlation to the estimated mean blood glucose is determined from studies in persons with normal erythrocyte turnover of approximately 120 days and without severe chronic kidney disease (CKD). Several smaller studies have shown that HbA1c in persons with type 2 diabetes and CKD, especially on chronic haemodialysis, is an uncertain marker of the mean blood glucose. Generally, studies show that HbA1c underestimate the actual mean blood glucose. The reason for a false low HbA1c in persons with type 2 diabetes and with CKD has yet to be established. However, it is known that erythropoietin treatment and iron infusion increases the erythropoiesis, which results in new non-glycated erythrocytes, and this is likely to lower HbA1c. The erythrocyte life span is found to be reduced in persons on dialysis, which in combination with blood loss from the dialysis also contributes to a reduction in HbA1c. The shorter erythrocyte life span is thought to be due to the toxic uraemic environment as well as mechanical damage caused by haemodialysis.

Objective:

To investigate the correlation between the mean glucose concentration measured by CGM and the estimated mean blood glucose from HbA1c in persons with type 2 diabetes and on chronic haemodialysis compared to a control groups of persons with type 2 diabetes and normal renal function.

Method:

Prospective case-control study over 17 weeks with 40 persons in each group. The case group consist of 40 persons with type 2 diabetes and on chronic haemodialysis. The control group consists of persons with type 2 diabetes and normal renal function (defined as and estimated glomerular filtration rate (eGFR) above 60 ml/min). CGM is performed for a maximum of seven days on week 0, 4, 8, 12 and 16 of the study period with simultaneous analysis of glycaemic markers (HbA1c, glycated albumine and fructosamine). Each of the first five visit was conducted with 3 to 5 weeks interval and the final visit not more than two weeks after the final visit. The erythrocyte life span will be measured with an isotope (Crom-51) method in both the dialysis group and the control group, to establish if diminished erythrocyte life span and falsely low HbA1c is correlated.

Statistical methods:

The null hypothesis is that there is no difference between the ratio of total mean glucose from CGM and estimated mean blood glucose from HbA1c at week 17 when measured in type 2 diabetic persons on chronic haemodialysis compared to type 2 diabetic persons with normal renal function.

The alternative hypothesis is that there is a difference in the ratio between the groups which in a pilot study of persons with diabetes on chronic haemodialysis was found to be 0.16 (mean glucose from CGM/mean blood glucose from HbA1c) when compared to persons with diabetes with out nephropathy.

From one of the pilot arms ώ = 0.148 and σ = 0.128 were extracted. The following scenarios were considered; β(0) = 0 and β (1) = 0, 0.01, ..., 0.2 and n = 40. For each scenario, 5000 data sets were simulated in accordance with the above specifications. Each data set was analyzed by a mixed linear model with treatment arm as fixed effect and person as random effect. The hypothesis β(0) = β(1) was tested at a significance of 5%. The simulated effect in each scenario was calculated as the fraction of rejections in the 5000 tests. Datasets were simulated in the statistical programming language R (www.r-project.org). The smallest difference in the ratio of mean glucose from CGM and mean blood glucose from HbA1c that could be detected with a power of 80% based on the likelihood ratio test described above and using a 5% significance level was 0.1 for n=40 per arm.

ELIGIBILITY:
Inclusion criteria for case group (on chronic haemodialysis with type 2 diabetes):

* Type 2 diabetes*
* BMI 17.5-50 kg/m2
* Receiving antidiabetic treatment
* Chronic haemodialysis treatment for a minimum of 3 months
* 24 hour urinary protein excretion of less than 10.0 g/day at screening or within the last 6 months

Exclusion criteria for case group (on chronic haemodialysis with type 2 diabetes):

* Type 1 diabetes
* Acute or chronic pancreatitis
* Intermittent treatment with steroid during study period (defined as more than two days)
* Haemoglobin < 6.0 mmol / l (day of screening)
* Hypertriglyceridemia (≥ 10mmol / L)
* Hyperbilirubinemia (≥ 35 μmol / L)
* Pregnant or breast-feeding
* Blood transfusion within the last 3 months
* Blood transfusion during the investigation period
* Splenectomy
* High alcohol consumption (defined as more than 21 units per week)
* Vitamin E supplement
* Ribavirin treatment
* Interferon Alpha treatment
* Positive for haemoglobinopathy (examined for haemoglobinopathy if patients come from Africa, Mediterranean, Middle East, Iran, Iraq, India, Pakistan or Southeast Asia)
* Severe infections

Inclusion criteria for control group (type 2 diabetes and normal renal function):

* Type 2 diabetes*
* BMI 17.5-50 kg / m2
* Receiving antidiabetic treatment
* Plasma creatinine in the normal range (men: 60-105 μmol/l, women: 45-90 μmol/l)
* eGFR > 60 ml/min/1.73m2
* Urinary Albumin-to-Creatinine Ratio < 300mg/g or 24h urinary protein excretion <0.3g at screening or within the last 6 months

Exclusion criteria for control group (type 2 diabetes and normal renal function):

* Type 1 diabetes
* Acute or chronic pancreatitis
* Intermittent treatment with steroid during study period (defined as more than two days)
* Haemoglobin <7.3 mmol / l for women
* Haemoglobin <8.3 mmol / l for men
* Hypertriglyceridemia (≥ 10mmol / L)
* Hyperbilirubinemia (≥ 35 μmol / L)
* Pregnant or breast-feeding
* Blood transfusion within the last 3 months
* Blood transfusion during the investigation period
* Splenectomy
* Intermittent treatment with steroid during study period (defined as more than two days)
* High alcohol consumption (defined as more than 21 units per week)
* Vitamin E supplement
* Ribavirin
* Interferon Alpha treatment
* Positive for haemoglobinopathy (examined for haemoglobinopathy if patients come from Africa, Mediterranean, Middle East, Iran, Iraq, India, Pakistan or Southeast Asia)
* Severe infections

  *Inclusion with diagnosis of type 2 diabetes was defined as ongoing antidiabetic treatment and previously diagnosed with type 2 diabetes according to the following criteria:
* A random venous plasma glucose concentration ≥ 11.1 mmol/l or
* A fasting plasma glucose concentration ≥ 7.0 mmol/l (whole blood ≥ 6.1 mmol/l) or
* Two hour plasma glucose concentration ≥ 11.1 mmol/l two hours after 75g anhydrous glucose in an oral glucose tolerance test or
* HbA1c above 48 mmol/mol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total of 80 participants with 40 patients in each group.
  Case group: 40 patients on chronic haemodialysis with type 2 diabetes.
  Control group: 40 patients with type 2 diabetes and normal renal function (defined as eGFR >60 ml/min and with urinary protein excretion below 0.3g/day (24 hour urine collection) or 300mg/g (Urinary Albumin-to-Creatinine Ratio).
  The patients are recruited from the department of Endocrinology or Nephrology at Rigshospitalet, from Herlev Hospital department of Nephrology, Gentofte Hospital and Steno Diabetes Center Copenhagen, Hillerød Hospital department of Endocrinology or Nephrology and Roskilde Hospital department of Nephrology.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
HbA1c evaluated by the total mean glucose from continuous glucose monitoring | 17 weeks
  Difference between groups in the ratio of total mean glucose measured by continuous glucose monitoring over the estimated mean blood glucose from HbA1c measured at week 17. For each CGM measurement at least 48 hours must be completed and three out of five periods with CGM. In total a least 14 days must be completed.

SECONDARY OUTCOMES:
Erythrocyte life span | 4 weeks
  Erythrocytes are labelled with Cr-51 and reinjected 3 hours after incubation. Blood samples for counts per minute will be taken twice a week the following four weeks which makes it possible to extrapolate the curve of the erythrocyte life span for each patient.
Glycated albumin | 17 weeks
  Plots illustrating the correlation between mean glucose from continuous glucose monitoring and glycated albumin (%) for each week
Fructosamine | 17 weeks
  Plots illustrating the correlation between mean glucose from continuous glucose monitoring and fructosamine (μmol/l) for each week
HbA1c evaluated by the mean glucose from continuous glucose monitoring for each week | 17 weeks
  Plots illustrating the correlation between mean glucose from continuous glucose monitoring and HbA1c for each week
Blood volume | 4 hours
  Carbon monoxide rebreathing method for measurements of total blood volume (liter), plasma volume (liter) and erythrocyte volume (liter)
Standard deviation | 17 weeks
  Standard deviation for glycaemic variability measured by continuous glucose monitoring in both Groups. For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Coefficient variation | 17 weeks
  Coefficient variation for glycaemic variability measured by continuous glucose monitoring in both groups. For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately. A coefficient variation below 36% is considered stable and above is considered unstable.
Low Blood Glucose Index | 17 weeks
  Low Blood Glucose Index for glycaemic variability measured by continuous glucose monitoring in both Groups. Is a risk index for predicting hypoglycaemia. For the group on haemodialysis the days of haemodialysis and days without haemodialysis will also be evaluated separately.
High Blood Glucose Index | 17 weeks
  High Blood Glucose Index for glycaemic variability measured by continuous glucose monitoring in both groups. Is a risk index for predicting hyperglycaemia. For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Time in hypoglycaemic range below 3.0 mmol/l | 17 weeks
  Time in hypoglycaemic range(%) below 3.0 mmol/l evaluated by continuous glucose monitoring . For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Time in hypoglycaemic range below 3.9 mmol/l to 3.0 mmol/l | 17 weeks
  Time in hypoglycaemic range(%) below 3.9 mmol/l to 3.0 mmol/l evaluated by continuous glucose monitoring . For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Time in target range from 3.9 mmol/l to 10.0 mmol/l | 17 weeks
  Time in target range(%) from 3.9 mmol/l to 10.0 mmol/l evaluated by continuous glucose monitoring . For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Time in hyperglycaemic range above 10.0 mmol/l | 17 weeks
  Time in hyperglycaemic range(%) above 10.0 mmol/l evaluated by continuous glucose monitoring . For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Time in hyperglycaemic range above 13.9 mmol/l | 17 weeks
  Time in hyperglycaemic range(%) above 13.9 mmol/l evaluated by continuous glucose monitoring . For the group on haemodialysis the days of haemodialysis and the days without haemodialysis will also be evaluated separately
Hypoglycaemic events | 17 weeks
  Beginning of a CGM event is defined as a reading below the threshold for at least 15 min for either a value below 3.0 mmol/l or between 3.9 mmol/l to 3.0 mmol/l. The end of a CGM event is defined as a reading for 15 min above 3.9 mmol/l.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Denmark